CLINICAL TRIAL: NCT01353677
Title: Pilot Study to Assess the Feasibility of Collecting Quality of Life Data in Collaboration With the Stem Cell Therapeutic Outcomes Database
Brief Title: Feasibility of Collecting Quality of Life Data in Collaboration With the Stem Cell Therapeutic Outcomes Database
Acronym: 09-SQOL
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: 09-SQOL
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic stem cell transplantation; QOL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HSCT recipients: 1. Adult (≥ 18 years), or pediatric (≥ 2 years and < 18 years) allogeneic HCT recipient (related, unrelated, or CBU) at participating pilot study transplant centers.
  2. Signed informed consent form from adult patient or parent/guardian of pediatric patient.
  3. Patient must have a valid mailing address within the United States to receive QOL surveys.
  4. Ability to speak and read English.
  5. Patients with access to a telephone.

SUMMARY:
This is a multi-institution, non-randomized, prospective pilot study to evaluate the feasibility of collecting quality of life (QOL) data on a large cohort of pediatric and adult allogeneic Hematopoietic stem cell transplantation (HCT) recipients.

DETAILED DESCRIPTION:
QOL data will be collected at baseline (pre-transplant), 100 days, 6 months, and 12 months post transplant. The transplant center will consent the patient and administer the baseline QOL surveys. The transplants center will then submit the competed baseline data and patient contact information to the Center for International Blood and Marrow Transplant Research (CIBMTR). The remaining surveys will be administered to the patient from the CIBMTR via paper surveys mailed to the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years), or pediatric (≥ 2 years and < 18 years) allogeneic HCT recipient (related, unrelated, or CBU) at participating pilot study transplant centers.
2. Signed informed consent form from adult patient or parent/guardian of pediatric patient.
3. Patient must have a valid mailing address within the United States to receive QOL surveys.
4. Ability to speak and read English.
5. Patients with access to a telephone.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult allogeneic HCT recipients
Sampling Method: Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2014-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Rizzo, MD, MS, Principal Investigator — CIBMTR/ Medical College of Wisconsin
Locations (7):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington